CLINICAL TRIAL: NCT05443893
Title: Application Research of Key Points Detection Technology of Artificial Intelligence in Kinematics Analysis
Brief Title: Artificial Intelligence in Kinematics Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhou Mouwang, Professor, Peking University Third Hospital
Other Study IDs: M2021231
Record Dates: First submitted 2022-06-03; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-07

CONDITIONS: Gait

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Normal subjects: Gait analysis with artificial intelligence and traditional methods
  Interventions: Device: Application Research of key points detection technology
- Subjects with abnormal gait: Gait analysis with artificial intelligence and traditional methods
  Interventions: Device: Application Research of key points detection technology

INTERVENTIONS:
Device: Application Research of key points detection technology — Artificial intelligence human key point detection model mainly has traditional algorithm, "top-down" algorithm and "bottom-up" algorithm three methods, three methods have advantages. This project will comprehensively use the above three methods to conduct algorithm and parameter debugging in the public data set and test in the private data set, so as to obtain the most suitable human key point recognition method for gait analysis

SUMMARY:
1. Establish data sets. The private data set includes relevant parameters including video of the subject's gait and standard methods for kinematic analysis;
2. Develop new models. Based on public and private data sets, the kinematic analysis model of human key point detection is further developed.
3. Test the new model. By comparing the parameters with the standard method, the accuracy of the model was verified, and the kinematics analysis model of artificial intelligence with accuracy above 98% was obtained

DETAILED DESCRIPTION:
Artificial intelligence human key point detection model mainly has traditional algorithm, "top-down" algorithm and "bottom-up" algorithm three methods, three methods have advantages. This project will comprehensively use the above three methods to conduct algorithm and parameter debugging in the public data set and test in the private data set, so as to obtain the most suitable human key point recognition method for gait analysis

ELIGIBILITY:
Inclusion Criteria:

* 1. Abnormal gait.
* Can walk 6m or more independently.
* Older than 18.

Exclusion Criteria:

* Fracture may be aggravated by walking in the acute stage or early postoperative stage. Have heart, lung, liver and kidney And other serious diseases, heart function grading greater than GRADE I (NYHA), respiratory failure and other symptoms and signs or Check the results.
* The mental and psychological state cannot cooperate with the completion of the experiment.
* High risk of falls (Berg score ≤20）
* Gait kinematics analysis equipment cannot be used together.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Normal gait subjects and abnormal gait subjects
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-07-10 (Estimated); Primary Completion 2022-07-29 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Gait related parameters | 30mins
  Step frequency/pace/gait cycle/step length